CLINICAL TRIAL: NCT05810363
Title: The Safety of Etomidate - Propofol Mixture vs Propofol in Total Intravenous Anesthesia During Abdominal Surgery : a Randomized, Double-blind, Controlled, Multicenter Study
Brief Title: The Safety of Etomidate - Propofol Mixture vs Propofol in Total Intravenous Anesthesia During Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ailin Luo (Other)
Responsible Party: Sponsor-Investigator, Ailin Luo, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEPT
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Etomidate; Hypotension
MeSH Terms: conditions — Hypotension | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EP group (Experimental): Patients in this group will receive etomidate- propofol mixture during induction and maintenance.
  Interventions: Drug: Etomidate - propofol mixture
- P group (Experimental): Patients in this group will receive propofol during induction and maintenance.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Etomidate - propofol mixture — Patients will receive etomidate - propofol mixture during induction and maintenance. Sufentanil 0.2-0.7 μg/kg，Cisatracurium 0.15 mg/kg，EP mixture（E：P=1:2） 0.1-0.25 ml/kg for induction, EP mixture 0.4~ 1.2 ml/kg/h and remifentanil 0.05μg/kg/min ~0.3 μg/kg/min for maintenance.
  Other Names: EP
  Arms: EP group
Drug: Propofol — Patients will receive propofol during induction and maintenance.Sufentanil 0.2-0.7 μg/kg，Cisatracurium 0.15 mg/kg，propofol 0.1-0.25 ml/kg for induction, propofol 0.4~ 1.2 ml/kg/h and remifentanil 0.05μg/kg/min ~0.3 μg/kg/min for maintenance.
  Other Names: P
  Arms: P group

SUMMARY:
The purpose of this study is to access the safety of etomidate - propofol mixture vs propofol in total intravenous anesthesia during abdominal surgery.

DETAILED DESCRIPTION:
Total intravenous anesthesia (TIVA) is one of the common anesthesia maintenance methods in clinic. Intravenous anesthetics commonly used in clinical practice include propofol and etomidate, both of which have their own advantages and disadvantages. Among them, propofol has the advantages of rapid onset, complete sedation and rapid recovery, but it is easy to cause injection pain. Moreover, the inhibitory effect of propofol on the circulatory system is more obvious, and the incidence of hypotension during propofol use in TIVA is higher. In contrast, intraoperative hypotension substantially increases the risk of perioperative adverse cardiovascular and cerebrovascular events. Etomidate, a derivative of imidazole, reversibly increases GABAA receptor activity and inhibits synaptic transmission and impulse transmission, resulting in sedation. Etomidate has a rapid onset of action, minimal hemodynamic effects, and a shorter dose-related half-life than propofol; however, etomidate has a suppressive effect on the adrenal cortex. Several studies have confirmed transient suppression of adrenocortical function with a single injection or continuous pump of etomidate, with recovery of preoperative baseline adrenocortical function within 48 hours after surgery.

Combined drugs can reduce the adverse reactions caused by single drugs. Considering the complementary effects of propofol and etomidate in pharmacodynamic characteristics, the combination of propofol and etomidate is beneficial to maximize their respective advantages and reduce adverse reactions.

Intraoperative hypotension is a common complication during general anesthesia, and severe hypotension is closely related to perioperative cardiovascular complications and stroke ; therefore, avoiding perioperative hypotension is the basic premise to ensure patient safety. Abdominal surgery is a common type of general surgery, with a large number of operations and relatively uniform operation time, which is easy to collect cases. Therefore, this study aims to investigate the effect of propofol-etomidate mixture used in TIVA on the incidence of hypotension during anesthesia induction and maintenance in adult patients undergoing elective abdominal surgery, in order to provide an alternative, safe, reasonable and easy to promote medication regimen for total intravenous anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA Ⅰ~Ⅲ;
* BMI was 18-28 kg/m2;
* For elective abdominal surgery under intravenous general anesthesia;
* The expected duration of anesthesia was 1 to 4 hours.

Exclusion Criteria:

* Pregnant patients;
* Septic shock and multiple organ failure diagnosed within 14 days;
* Hyperkalemia (serum potassium >5.5mmol/L) within 48 hours;
* Stroke or transient ischemic attack within 3 months;
* Patients with unstable angina pectoris or myocardial infarction within 3 months; Arrhythmia requiring treatment was not treated or treatment did not meet expectations;
* Patients with preoperative diagnosed diabetes mellitus and uncontrolled blood glucose; Diabetic complications were diagnosed before surgery, including diabetic ketoacidosis, hyperosmolar coma, diabetes-related infection, diabetic nephropathy, retinopathy, diabetic cardiomyopathy, diabetic neuropathy, diabetic foot, etc.
* Severe liver and renal dysfunction;
* Liver surgery, renal surgery, adrenal surgery, day surgery;
* Resting blood pressure ≥180/110 mmHg (2020 ISH hypertension guideline ≥ grade 3 hypertension); Or systolic blood pressure <90mmHg or mean blood pressure <65mmHg.
* Taking corticosteroids or other immunosuppressants for more than 10 days within 6 months or having a history of adrenal cortex suppression or immune system diseases;
* Patients who participated in other drug trials within 3 months;
* Patients with disturbance of consciousness or other mental diseases;
* Confirmed/suspected abuse or long-term use of narcotic sedatives and analgesics；
* Patients with cancer who received neoadjuvant therapy or chemotherapy before surgery;
* Allergic to the drug used in this trial and its components.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Incidence and duration of hypotension during anesthesia | during anesthesia
  Systolic blood pressure ≤90 mmHg, or > 20% reduction from baseline, or mean arterial pressure <65 mmHg, from the time when anesthesia induction began to the time before the patient complied with transfer out of PACU

SECONDARY OUTCOMES:
Success rate of sedation | during anesthesia
  ① Successful induction of anesthesia, MOAA/S score to 0 or BIS<60 within 3 minutes after the end of administration; ② During the maintenance of anesthesia, there was no single BIS>60 for more than 5 minutes or the cumulative BIS>60 for more than 20% of the anesthesia time, no anticipated limb movement, and no anesthesia rescue measures during the maintenance period
Recovery time | during anesthesia
  Time from drug withdrawal to extubation
The type and dosage of vasoactive drugs used during operation | during anesthesia
  The type and dosage of vasoactive drugs used during operation
The incidence of postoperative nausea and vomiting | 72 hours after surgery
  The incidence of postoperative nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Ailin Luo, Dr, Principal Investigator — Department of Anesthesiology of Tongji Hospital
Locations (1):
- Tongji hospital, Wuhan, China

IPD SHARING:
Plan to Share IPD: No